CLINICAL TRIAL: NCT00703794
Title: ev3 Researching AXIUM Coiling Experience and Recanalization (RACER)
Brief Title: Researching AXIUM Coiling Experience and Recanalization (RACER)
Acronym: RACER
Status: Completed | Type: Observational
Sponsor: Medtronic Neurovascular Clinical Affairs (Industry)
Responsible Party: Sponsor
Other Study IDs: ev3-FD1942-CR00045
Record Dates: First submitted 2008-06-23; First posted 2008-06-24 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Aneurysms; Vascular Diseases; Cerebrovascular Disorders; Intracranial Arterial Diseases
Keywords: ev3 Neurovascular; aneurysms; cerebrovascular; endovascular; neurovascular therapies; RACER; AXIUM; The AXIUM Progressive Coil System; ev3; MTI; Micro Therapeutics; FX detachable coil system; K060747; brain diseases
MeSH Terms: conditions — Aneurysm; Vascular Diseases; Cerebrovascular Disorders; Intracranial Arterial Diseases; Brain Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- AXIUM Coils
  Interventions: Device: The AXIUM Progressive Coil System

INTERVENTIONS:
Device: The AXIUM Progressive Coil System — Embolization of aneurysm

SUMMARY:
The data collected in this study will be used to support International Regulatory submissions. The study objective is to evaluate the continued safety and efficacy of the AXIUM Progressive Coil System.

This Device has been used clinically at approximately 150 Institutions under FDA 510(k) clearance since April 24, 2007. The device received CE authorization on June 30, 2007. Through December 2007, more than 1000 patients have been treated with the AXIUM Coils.

ELIGIBILITY:
Inclusion Criteria:

* Patient or patient's legally authorized representative has signed and dated an Informed Consent Form
* Must be at least 18 years of age
* Aneurysm location, angio-architecture, morphology, or medical condition, is considered by the neurosurgical / interventional team to be at very high risk for management by traditional operative techniques, or aneurysm is considered to be inoperable
* Patient is willing to conduct follow-up visits

Exclusion Criteria:

* Aneurysm was previously treated
* Patient has a cerebral aneurysm with a location, angioarchitecture or morphology that presents an unacceptable risk of morbidity due to the Study procedures
* Patient is participating in another clinical research Study
* Patient has a medical, social or psychological condition, which precludes the patient from receiving Study required treatment, evaluation, procedures and follow-up
* Female patient is pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intracranial aneurysm, either ruptured or un-ruptured, with aneurysm has a maximum diameter of 2mm to 20mm
Sampling Method: Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2008-06; Primary Completion 2012-01-16 (Actual); Study Completion 2012-01-16 (Actual)

PRIMARY OUTCOMES:
Percent Occlusion | Defined in protocol

SECONDARY OUTCOMES:
Morbidity/Mortality | Defined in protocol

CONTACTS AND LOCATIONS:
Overall Officials: Ajay K Wakhloo, MD, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (18):
- United States (18):
  - Lac+Usc/Uscuh, Los Angeles, California
  - Vascular and Interventional Specialists of Orange County, Inc. - St. Joseph Hospital of Orange, Orange, California
  - Lee Memorial Health System, Fort Myers, Florida
  - University of Miami - Jackson Memorial Hospital Systems, Miami, Florida
  - Bayfront Medical Center, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Neurologic & Orthopedic Hospital of Chicago (NOHC), Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - Abbott Northwestern, Minneapolis, Minnesota
  - Kaleida Health - Millard Fillmore, Buffalo, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Palmetto Richland Health Memorial Hospital, Columbia, South Carolina
  - Fletcher Allen Health Care, Burlington, Vermont
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Background] Casasco AE, Aymard A, Gobin YP, Houdart E, Rogopoulos A, George B, Hodes JE, Cophignon J, Merland JJ. Selective endovascular treatment of 71 intracranial aneurysms with platinum coils. J Neurosurg. 1993 Jul;79(1):3-10. doi: 10.3171/jns.1993.79.1.0003. PMID 8315465
- [Background] Wakhloo AK, Gounis MJ, Sandhu JS, Akkawi N, Schenck AE, Linfante I. Complex-shaped platinum coils for brain aneurysms: higher packing density, improved biomechanical stability, and midterm angiographic outcome. AJNR Am J Neuroradiol. 2007 Aug;28(7):1395-400. doi: 10.3174/ajnr.A0542. PMID 17698550
- [Background] Linfante I, Wakhloo AK. Brain aneurysms and arteriovenous malformations: advancements and emerging treatments in endovascular embolization. Stroke. 2007 Apr;38(4):1411-7. doi: 10.1161/01.STR.0000259824.10732.bb. Epub 2007 Feb 22. PMID 17322071
- [Background] Razack N, Thompson BG. Treatment of intracranial aneurysms: clipping or coiling? J Neuroophthalmol. 2004 Mar;24(1):1-2. doi: 10.1097/00041327-200403000-00001. No abstract available. PMID 15206430
- [Background] Mericle RA, Reig AS, Burry MV, Eskioglu E, Firment CS, Santra S. Endovascular surgery for proximal posterior inferior cerebellar artery aneurysms: an analysis of Glasgow Outcome Score by Hunt-Hess grades. Neurosurgery. 2006 Apr;58(4):619-25; discussion 619-25. doi: 10.1227/01.NEU.0000204127.81249.28. PMID 16575325
- [Background] Thornton J, Debrun GM, Aletich VA, Bashir Q, Charbel FT, Ausman J. Follow-up angiography of intracranial aneurysms treated with endovascular placement of Guglielmi detachable coils. Neurosurgery. 2002 Feb;50(2):239-49; discussion 249-50. doi: 10.1097/00006123-200202000-00003. PMID 11844258
- See also: ev3 Inc. — http://www.ev3.net